CLINICAL TRIAL: NCT02253953
Title: An Open Study to Investigate the Effect of Two Times Oral 100 mg Ritonavir Capsules on Pharmacokinetics of Single Doses of BILR 355 BS (Dose Steps: 5 and 12.5 mg) Dissolved in 5 mL PEG 400 After Oral Administration in Healthy Male Volunteers, and a Double Blind, Placebo Controlled Study for Doses From 25 mg to 100 mg BILR 355 BS
Brief Title: Pharmacokinetics of Single Doses of BILR 355 BS Given With Ritonavir in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1188.4
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ritonavir

ARMS (10):
- D1 (Experimental)
  Interventions: Drug: BILR 355 BS, D1; Drug: Ritonavir
- D2 (Experimental)
  Interventions: Drug: BILR 355 BS, D2; Drug: Ritonavir
- D3 (Experimental)
  Interventions: Drug: BILR 355 BS, D3; Drug: Ritonavir
- D4 (Experimental)
  Interventions: Drug: BILR 355 BS, D4; Drug: Ritonavir
- D5 (Experimental)
  Interventions: Drug: BILR 355 BS, D5; Drug: Ritonavir
- D6 (Experimental)
  Interventions: Drug: BILR 355 BS, D6; Drug: Ritonavir
- D7 (Experimental)
  Interventions: Drug: BILR 355 BS, D7; Drug: Ritonavir
- D8 (Experimental)
  Interventions: Drug: BILR 355 BS, D8; Drug: Ritonavir
- D10 (Experimental)
  Interventions: Drug: BILR 355 BS, D10; Other: high-fat breakfast; Drug: Ritonavir
- Placebo (Placebo Comparator): for D3 - D10
  Interventions: Drug: Placebo; Drug: Ritonavir

INTERVENTIONS:
Drug: BILR 355 BS, D1
  Arms: D1
Drug: BILR 355 BS, D2
  Arms: D2
Drug: BILR 355 BS, D3
  Arms: D3
Drug: BILR 355 BS, D4
  Arms: D4
Drug: BILR 355 BS, D5
  Arms: D5
Drug: BILR 355 BS, D6
  Arms: D6
Drug: BILR 355 BS, D7
  Arms: D7
Drug: BILR 355 BS, D8
  Arms: D8
Drug: BILR 355 BS, D10
  Arms: D10
Drug: Placebo
  Arms: Placebo
Other: high-fat breakfast
  Arms: D10
Drug: Ritonavir

SUMMARY:
Assessment of the effect of two times oral 100 mg ritonavir capsules on pharmacokinetics of a single dose of BILR 355 BS dissolved in PEG 400

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy males
* Age range from 21 to 50 years
* Body mass index (BMI) be within 18.5 to 29.9 kg/m2
* In accordance with Good Clinical Practice and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial

Following exclusion criteria are of special interest for this study:

* Erythema, exanthema and comparable skin alterations

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2002-11; Primary Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration of the analyte in plasma (Cmax) | up to 120 hours after drug administration
Time to reach Cmax (tmax) | up to 120 hours after drug administration
Area under the concentration-time curve (AUC) | up to 120 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 120 hours after drug administration
Total clearance of the analyte in plasma (CL/F) | up to 120 hours after drug administration
Total mean residence time (MRTtot) | up to 120 hours after drug administration
Apparent volume of distribution (Vz/F) | up to 120 hours after drug administration
Renal clearance (CLR) | up to 72 hours after drug administration
Urinary excretion (Ae) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 26 days